CLINICAL TRIAL: NCT05267106
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib in Participants With Previously Treated Glioblastoma or Other Primary Central Nervous System Tumors Harboring Activating FGFR1-3 Alterations (FIGHT-209)
Brief Title: Study to Evaluate the Efficacy and Safety of Pemigatinib in Participants With Previously Treated Glioblastoma or Other Primary Central Nervous System Tumors Harboring Activating FGFR1-3 Alterations
Acronym: FIGHT-209
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment ceased after a pre-planned futility interim analysis indicated a low probability to confer a clinically meaningful improvement in objective response when compared to currently available therapies. There were no safety related concerns.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-209; 2021-004740-24 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-03-04 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma; Adult-type Diffuse Gliomas
Keywords: glioblastoma; GBM; adult-type diffuse gliomas; gliomas; oligodendroglioma; FGFR1-3 Alteration; FGFR1-3 fusions; FGFR1-3 rearrangements; Central nervous system tumor; isocitrate dehydrogenase; IDH-mutant astocytoma; IDH-wild-type GBM; glioneuronal; neuronal; circumscribed astrocytic glioma
MeSH Terms: conditions — Glioblastoma; Glioma; Oligodendroglioma; Central Nervous System Neoplasms | interventions — pemigatinib

STUDY DESIGN:
Intervention Model Description: This study consists of 2 cohorts and participants will receive pemigatinib 13.5 mg QD on a 2-week on-therapy and 1-week off-therapy schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: IDH-wild-type GBM (Experimental): Participants with histopathologically proven, WHO Grade 4, IDH-wild-type GBM OR molecular diagnosis of IDH-wild-type, diffuse astrocytic glioma with molecular features of Grade 4 GBM that are recurrent, harboring FGFR1-3 fusions/or other rearrangements, or with a defined FGFR1-3 mutation or in-frame deletion.
  Interventions: Drug: Pemigatinib
- Cohort B: Other gliomas other than GBM (Experimental): Participants with other histopathologically proven gliomas other than GBM, circumscribed astrocytic gliomas, and glioneuronal and neuronal tumors that are recurrent, harboring FGFR1-3 fusions/or other rearrangements or with a defined FGFR1-3 activating mutation or in-frame deletion
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — 13.5mg tablet taken every morning (unless otherwise directed) for 2 weeks and then 1 week off.
  Other Names: NCB054828

SUMMARY:
This is an open-label, monotherapy study of pemigatinib in participants with recurrent glioblastoma (GBM) or other recurrent gliomas, circumscribed astrocytic gliomas, and glioneuronal and neuronal tumors with an activating FGFR1-3 mutation or fusion/rearrangement. This study consists of 2 cohorts, Cohorts A, and B, and will enroll approximately 82 participants into each cohort. Participants will receive pemigatinib 13.5 mg QD on a 2-week on-therapy and 1-week off-therapy schedule as long as they are receiving benefit and have not met any criteria for study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Histological, cytological, or molecular confirmation of recurrent GBM or other glioma, circumscribed astrocytic glioma, or glioneuronalor neuronal tumors that has recurred.
* Radiographically measurable disease.

  . -Karnofsky performance status ≥ 60.
* Life expectancy ≥ 12 weeks.
* Documentation of an actionable FGFR1-3 gene mutation or fusion/rearrangement from tissue : FGFR1-3 fusions or other rearrangements (FGFR1-3 in-frame fusions, any FGFR2 rearrangement, or FGFR1/3 rearrangement with known partner) or a defined FGFR1-3 activating mutation or in-frame deletion. Only participants with FGFR fusions or rearrangements with an intact kinase domain are eligible.
* MRI-documented objective progression after prior therapy and must have no therapy available that is likely to provide clinical benefit.
* Most recent archival tumor specimen must be a tumor block or a minimum of 15 unstained slides from biopsy or resection of primary tumor or metastasis.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Prior receipt of an FGFR inhibitor.
* Receipt of anticancer medications or investigational drugs for any indication or reason within 28 days before first dose of study drug.
* Participants may have had treatment for an unlimited number of prior relapses but must not have had prior bevacizumab or other VEGF/VEGFR inhibitors (exception: prior bevacizumab is allowed if it was administered for the treatment of radiation necrosis rather than progressive tumor and was stopped at least 12 weeks prior to MRI showing tumor progression).
* Concurrent anticancer therapy
* Candidate for potentially curative surgery.
* Dexamethasone (or equivalent) > 4 mg daily at the time of study registration
* Current evidence of clinically significant corneal or retinal disorder as confirmed by ophthalmologic examination.
* Diffuse leptomeningeal disease.
* Radiation therapy administered within 12 weeks before enrollment/first dose of study drug.
* Known additional malignancy that is progressing or requires active systemic treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ebiana, MD, Study Director — Incyte Corporation
Locations (79):
- United States (32):
  - Valkyrie Clinical Trials, Beverly Hills, California
  - City of Hope National Medical Center, Duarte, California
  - Providence Medical Foundation, Fullerton, California
  - Usc Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Neuroscience Health Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Providence St Joseph Hospital Orange Center For Cancer Prevention and Treatment, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Baptist Md Anderson Cancer Center, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute Downtown Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Tampa, Florida
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Minnesota Health Clinics and Surgery Center, Minneapolis, Minnesota
  - Northwell Health, Lake Success, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - UC Health At Cincinnati Va Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Denmark (3):
  - Aalborg Universitets Hospital, Aalborg
  - Rigshospitalet Uni of Hospital of Copenhagen, Copenhagen
  - Odense University Hospital, Odense C
- France (4):
  - Chru de Lille Hopital Claude Huriez, Lille
  - Chu Hopital de La Timone, Marseille
  - Hospital Universitaire Pitie-Salpetriere, Paris
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
- Germany (4):
  - Universitatsklinikum Bonn Aoer, Bonn
  - Klinikum Der Johann Wolfgang Goethe University, Frankfurt
  - Universitaetsklinikum Heidelberg, Heidelberg
  - University Hospital Tuebingen, Tübingen
- Italy (6):
  - Ospedale Bellaria, Bologna
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - A.S.L. Napoli 1 Centro Ospedale Del Mare, Ponticelli
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliero Universitaria Citta Della Salute E Della Scienza, Torino
- Japan (6):
  - University of Tokyo Hospital, Bunkyō City
  - National Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Nagoya University Hospital, Nagoya
  - Tohoku University Hospital, Sendai
- Netherlands (2):
  - Netherlands Cancer Institute Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus Mc Cancer Institute, Rotterdam
- Spain (14):
  - Hospital Del Mar, Barcelona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic Barcelona Main, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Ico Girona Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Ico Institut Catala D Oncologia, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (8):
  - Addenbrooke'S Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - St James'S University Hospital, Leeds
  - Guys Hospital, London
  - The Royal Marsden Nhs Foundation Trust - Sutton, London
  - The Royal Marsden Nhs Foundation Trust - Chelsea, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 31 study centers in Denmark, France, Germany, Italy, Japan, Netherlands, Spain, the United Kingdom, and the United States.
Groups:
- Recurrent Glioblastoma: Participants with recurrent glioblastoma with defined activating fibroblast growth factor receptor (FGFR) gene alterations received pemigatinib 13.5 milligrams (mg) once daily (QD) on a 2-week on-therapy and 1-week off-therapy schedule as long as they were receiving benefit and had not met any criteria for treatment discontinuation. Defined activating gene alterations included FGFR 1-3 fusions or rearrangements with intact FGFR kinase domain, or a defined set of FGFR 1-3 activating mutations or in-frame deletions.
- Recurrent Non-glioblastoma CNS Tumors: Participants with recurrent non-glioblastoma central nervous system (CNS) tumors with defined activating FGFR gene alterations received pemigatinib 13.5 milligrams (mg) once daily (QD) on a 2-week on-therapy and 1-week off-therapy schedule as long as they were receiving benefit and had not met any criteria for treatment discontinuation. Defined activating gene alterations included FGFR 1-3 fusions or rearrangements with intact FGFR kinase domain, or a defined set of FGFR 1-3 activating mutations or in-frame deletions.
Period: Overall Study
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Started | 74 | 9
Completed | 0 | 0
Not Completed | 74 | 9
Not completed — Death | 50 | 2
Not completed — Study terminated by Sponsor | 24 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors | Total
Number analyzed (Participants) | 74 | 9 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.45) | 39.2 (12.75) | 55.1 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 3 | 33
  Male | 44 | 6 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 60 | 6 | 66
  Unknown or Not Reported | 13 | 3 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 58 | 6 | 64
  Black/African-American | 2 | 0 | 2
  Asian | 2 | 0 | 2
  Not Reported | 7 | 1 | 8
  Unknown | 5 | 1 | 6
  Captured as "Other" in Database | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Participants With Recurrent Glioblastoma Based on Independent Central Review
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete response (CR) or partial response (PR) based on Response Assessment in Neuro-Oncology (RANO) as determined by an independent centralized radiological review committee. CR requires all of the following: disappearance of all enhancing measurable/nonmeasurable disease sustained for ≥4 weeks; no new lesions; stable/improved nonenhancing lesions; off corticosteroids/on physiologic replacement doses only and stable/improved clinically. PR requires all of the following: ≥50% decrease, compared with baseline, in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for ≥4 weeks; no progression of nonmeasurable disease; no new lesions; stable or improved nonenhancing lesions on same/lower dose of corticosteroids compared with baseline scan; on a corticosteroid dose not greater than the dose at time of baseline scan and stable/improved clinically.
Time Frame: up to 651 days
Population: Full Analysis Set: all enrolled participants who received at least 1 dose of pemigatinib. The 95% confidence interval (CI) was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 0
percentage of participants
  Confirmed tumor responses | 5.4 [1.49 to 13.27] |
  Unconfirmed tumor responses | 8.1 [3.03 to 16.82] |

2. Secondary Outcome: ORR in Participants With Recurrent Non-glioblastoma Central Nervous System Tumors Based on Independent Central Review
Description: ORR was defined as the percentage of participants who achieved a best overall response of CR or PR based on RANO as determined by an independent centralized radiological review committee. CR requires all of the following: disappearance of all enhancing measurable/nonmeasurable disease sustained for ≥4 weeks; no new lesions; stable/improved nonenhancing lesions; off corticosteroids/on physiologic replacement doses only and stable/improved clinically. PR requires all of the following: ≥50% decrease, compared with baseline, in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for ≥4 weeks; no progression of nonmeasurable disease; no new lesions; stable or improved nonenhancing lesions on same/lower dose of corticosteroids compared with baseline scan; on a corticosteroid dose not greater than the dose at time of baseline scan and stable/improved clinically.
Time Frame: up to 784 days
Population: Full Analysis Set. The 95% CI was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 0 | 9
percentage of participants
  Confirmed tumor responses |  | 22.2 [2.81 to 60.01]
  Unconfirmed tumor responses |  | 22.2 [2.81 to 60.01]

3. Secondary Outcome: Duration of Confirmed Response Based on Independent Central Review
Description: Duration of response was defined as the time from the first assessment of confirmed CR or PR until progressive disease (PD) (according to RANO and assessed by an independent centralized radiological review committee) or death (whichever occurred first). Progression was defined by any of the following: ≥25% increase in the sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of nonmeasurable lesions; or definite clinical deterioration not attributable to other causes apart from the tumor, or to decrease in corticosteroid dose.
Time Frame: up to 784 days
Population: Full Analysis Set. Only those participants with a confirmed CR or PR were analyzed. The 95% CIs were calculated using the Brookmeyer and Crowley method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 4 | 2
months | NA [NA to NA] — The median and the lower and upper bounds of the confidence interval were not estimable because no responders had disease progression or died. | NA [NA to NA] — The median and the lower and upper bounds of the confidence interval were not estimable because no responders had disease progression or died.

4. Secondary Outcome: Duration of Unconfirmed Response Based on Independent Central Review
Description: Duration of response was defined as the time from the first assessment of unconfirmed CR or PR until progressive disease (PD) (according to RANO and assessed by an independent centralized radiological review committee) or death (whichever occurred first). Progression was defined by any of the following: ≥25% increase in the sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of nonmeasurable lesions; or definite clinical deterioration not attributable to other causes apart from the tumor, or to decrease in corticosteroid dose.
Time Frame: up to 784 days
Population: Full Analysis Set. Only those participants with an unconfirmed CR or PR were analyzed. The 95% CIs were calculated using the Brookmeyer and Crowley method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 6 | 2
months | NA [1.74 to NA] — The median and the upper bound of the confidence interval were not estimable because too few responders had disease progression or died. | NA [NA to NA] — The median and the lower and upper bounds of the confidence interval were not estimable because no responders had disease progression or died.

5. Secondary Outcome: ORR as Determined by Investigator Assessment
Description: ORR was defined as the percentage of participants who achieved an unconfirmed best overall response of CR or PR based on RANO as determined by investigator assessment. CR requires all of the following: disappearance of all enhancing measurable/nonmeasurable disease sustained for ≥4 weeks; no new lesions; stable/improved nonenhancing lesions; off corticosteroids/on physiologic replacement doses only and stable/improved clinically. PR requires all of the following: ≥50% decrease, compared with baseline, in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for ≥4 weeks; no progression of nonmeasurable disease; no new lesions; stable or improved nonenhancing lesions on same/lower dose of corticosteroids compared with baseline scan; on a corticosteroid dose not greater than the dose at time of baseline scan and stable/improved clinically.
Time Frame: up to 784 days
Population: Full Analysis Set. The 95% CIs were calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
percentage of participants | 8.1 [3.03 to 16.82] | 22.2 [2.81 to 60.01]

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE reported for the first time or the worsening of a pre-existing event after the first dose of pemigatinib and within 30 days of the last dose of pemigatinib.
Time Frame: up to 814 days
Population: Safety Population: all enrolled participants who received at least 1 dose of pemigatinib
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
Participants | 73 | 9

7. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. A TEAE was defined as an AE reported for the first time or the worsening of a pre-existing event after the first dose of pemigatinib and within 30 days of the last dose of pemigatinib. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 814 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
Participants | 27 | 3

8. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation of Pemigatinib, Pemigatinib Dose Interruption, and Pemigatinib Dose Reduction
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as an AE reported for the first time or the worsening of a pre-existing event after the first dose of pemigatinib and within 30 days of the last dose of pemigatinib.
Time Frame: up to 814 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
Participants
  TEAEs leading to discontinuation of pemigatinib | 2 | 0
  TEAEs leading to pemigatinib dose interruption | 22 | 4
  TEAEs leading to pemigatinib dose reduction | 5 | 2

9. Secondary Outcome: Disease Control Rate (DCR) Based on Independent Central Review
Description: DCR was defined as the percentage of participants who achieved a best overall response of CR, PR, or stable disease (SD) based on RANO as determined by an independent centralized radiological review committee. In the case of SD, measurements must have met the SD criteria after the date of the first dose at a minimum interval of 42 days. SD occurred if the participant didn't qualify for CR, PR, or PD and required the following: stable nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan and clinically stable status.
Time Frame: up to 784 days
Population: Full Analysis Set. The 95% CIs were calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
percentage of participants
  Confirmed tumor responses | 36.5 [25.60 to 48.49] | 66.7 [29.93 to 92.51]
  Unconfirmed tumor responses | 36.5 [25.60 to 48.49] | 66.7 [29.93 to 92.51]

10. Secondary Outcome: Progression-free Survival (PFS) Based on Independent Central Review
Description: PFS was defined as the time from the first dose until progressive disease (according to RANO and assessed by an independent centralized radiological review committee) or death (whichever occurred first). Progression was defined by any of the following: ≥25% increase in the sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of nonmeasurable lesions; or definite clinical deterioration not attributable to other causes apart from the tumor, or to decrease in corticosteroid dose.
Time Frame: up to 784 days
Population: Full Analysis Set. The 95% CIs were calculated using the Brookmeyer and Crowley method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
months | 2.07 [2.04 to 2.37] | NA [1.74 to NA] — The median and the upper bound of the confidence interval were not estimable because too few participants had disease progression or died.

11. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first dose of study drug to death due to any cause.
Time Frame: up to 784 days
Population: Full Analysis Set. The 95% CIs were calculated using the Brookmeyer and Crowley method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors
Number analyzed (Participants) | 74 | 9
months | 11.37 [9.23 to 14.85] | 24.08 [18.79 to NA] — The upper bound of the confidence interval was not estimable because too few participants died.

ADVERSE EVENTS:
Time Frame: up to 814 days
Description: Adverse events have been reported for the Safety Population, comprised of all enrolled participants who received at least 1 dose of pemigatinib.
Groups:
- Total: Total
Arm/Group | Recurrent Glioblastoma | Recurrent Non-glioblastoma CNS Tumors | Total
All-Cause Mortality (participants affected / at risk) | 50/74 | 2/9 | 52/83
Serious Adverse Events (participants affected / at risk) | 17/74 | 0/9 | 17/83
Other Adverse Events (participants affected / at risk) | 71/74 | 9/9 | 80/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent Glioblastoma (N=74) | Recurrent Non-glioblastoma CNS Tumors (N=9) | Total (N=83)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Stroke-like migraine attacks after radiation therapy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent Glioblastoma (N=74) | Recurrent Non-glioblastoma CNS Tumors (N=9) | Total (N=83)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 1 (1) | 6 (8)
Alanine aminotransferase increased (Investigations) | 12 (15) | 2 (3) | 14 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (16) | 7 (9) | 23 (25)
Amylase decreased (Investigations) | 0 (0) | 1 (4) | 1 (4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Aphasia (Nervous system disorders) | 7 (7) | 0 (0) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (3) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 2 (3) | 6 (8)
Asthenia (General disorders) | 10 (17) | 2 (3) | 12 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Blood creatinine increased (Investigations) | 5 (5) | 2 (2) | 7 (7)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood parathyroid hormone decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood phosphorus increased (Investigations) | 5 (5) | 1 (1) | 6 (6)
Blood urea decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Chalazion (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
Confusional state (Psychiatric disorders) | 6 (7) | 0 (0) | 6 (7)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 16 (17) | 4 (4) | 20 (21)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 3 (3)
Cortisol decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 4 (4)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 33 (57) | 8 (12) | 41 (69)
Dry eye (Eye disorders) | 8 (9) | 3 (3) | 11 (12)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 3 (4) | 13 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (14) | 5 (5) | 16 (19)
Dysgeusia (Nervous system disorders) | 8 (8) | 2 (2) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Eyelash thickening (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (8) | 0 (0) | 6 (8)
Fatigue (General disorders) | 21 (23) | 3 (3) | 24 (26)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Gonadotrophin deficiency (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1) | 4 (4)
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 14 (16) | 1 (4) | 15 (20)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4) | 2 (4) | 4 (8)
Hyperphosphataemia (Metabolism and nutrition disorders) | 54 (89) | 7 (11) | 61 (100)
Hypertension (Vascular disorders) | 5 (6) | 0 (0) | 5 (6)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (7) | 0 (0) | 5 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 16 (21) | 4 (6) | 20 (27)
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 4 (4)
Keratopathy (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Lipase decreased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Lipase increased (Investigations) | 5 (7) | 1 (5) | 6 (12)
Lymphocyte count decreased (Investigations) | 4 (5) | 0 (0) | 4 (5)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 15 (15) | 1 (1) | 16 (16)
Nail infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9) | 2 (2) | 11 (11)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 4 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Onycholysis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 8 (8)
Onychomadesis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 5 (5)
Oral pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 4 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (8) | 0 (0) | 5 (8)
Paraesthesia (Nervous system disorders) | 5 (5) | 1 (1) | 6 (6)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (2) | 1 (1) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Punctate keratitis (Eye disorders) | 4 (5) | 0 (0) | 4 (5)
Pyrexia (General disorders) | 5 (6) | 1 (1) | 6 (7)
Retinal exudates (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
Seizure (Nervous system disorders) | 10 (13) | 1 (2) | 11 (15)
Skin infection (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 14 (21) | 0 (0) | 14 (21)
Taste disorder (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4)
Temperature regulation disorder (General disorders) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Vision blurred (Eye disorders) | 5 (5) | 1 (1) | 6 (6)
Vitamin D decreased (Investigations) | 4 (4) | 0 (0) | 4 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 5 (5) | 0 (0) | 5 (5)
White blood cell count decreased (Investigations) | 3 (5) | 1 (1) | 4 (6)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor after the prespecified interim analysis did not meet the futility boundary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT05267106/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT05267106/SAP_001.pdf